CLINICAL TRIAL: NCT06821087
Title: Evaluating the Neuromodulatory Effect of Ketamine in Long COVID: A Pilot Study Targeting Fatigue and Neurocognitive Symptoms
Brief Title: Evaluating the Neuromodulatory Effect of Ketamine in Long COVID-19
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Roots Behavioral Health (Unknown)
Responsible Party: Principal Investigator, William Michael Brode, Assistant Professor of Internal Medicine, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006367
Record Dates: First submitted 2025-02-10; First posted 2025-02-11 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Long COVID
Keywords: Long COVID; Post-COVID Condition; Post-Acute Sequelae of COVID-19; Brain Fog; Fatigue; Ketamine
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Mental Fatigue; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketamine Therapy (Experimental): Participants in this arm will receive four intramuscular (IM) ketamine injections over a two-week period. The initial dose will be 0.5 mg/kg during the first session, increasing to 0.65 mg/kg in the second session, and 0.75 mg/kg for the third and fourth sessions. Injections will be administered at least three days apart. All treatments will be conducted under medical supervision at a specialized clinic with standard safety protocols in place. Vital signs will be monitored before, during, and after each session to assess tolerability. Participants will also undergo assessments of fatigue, cognitive function, quality of life, and biomarkers pre- and post-treatment. Participants will receive fMRI imaging pre- and post-treatment.
  Interventions: Drug: Ketamine only

INTERVENTIONS:
Drug: Ketamine only — Participants in this arm will receive four intramuscular (IM) ketamine injections over a two-week period. The initial dose will be 0.5 mg/kg during the first session, increasing to 0.65 mg/kg in the second session, and 0.75 mg/kg for the third and fourth sessions. Injections will be administered at least three days apart.

SUMMARY:
Plain Language Summary:

This study is a clinical trial to see if ketamine can help treat symptoms of Long COVID, especially fatigue and problems with thinking clearly (often called "brain fog"). Long COVID is a condition that affects people even after they have recovered from COVID-19, causing ongoing health issues like tiredness, memory problems, and difficulty concentrating. Right now, there are very few treatments available for these symptoms, and many people are looking for new options to feel better.

What is the study trying to find out? Does ketamine help reduce fatigue and improve thinking skills in people with Long COVID? Does ketamine improve overall quality of life and mental health for people with Long COVID? Is ketamine safe and well-tolerated for people with Long COVID? How does ketamine affect the body's biological processes, like inflammation and brain function? How will the study work?

The study will include 20 adults between 18 and 65 years old who have Long COVID symptoms like fatigue or brain fog.

Participants will first meet with researchers to answer health questions, take surveys about their symptoms, and do tests to check their thinking skills. All participants will also have a brain scan (MRI) and give a blood sample to look at markers of inflammation.

Participants will then receive four ketamine treatments over two weeks at a specialized clinic. The ketamine will be given as an injection, with the dose slightly increasing during the treatment period.

After six weeks, participants will return for follow-up tests to see if their symptoms have improved. This includes repeating the surveys, thinking tests, MRI and blood test.

Why ketamine? Ketamine is a medicine originally used for anesthesia but has also been found to help with depression and other mental health issues. Researchers think it might help with Long COVID symptoms because it can reduce inflammation in the brain and improve how the brain functions. People with Long COVID often have signs of inflammation and changes in brain chemicals, which ketamine might help balance.

What are the potential benefits? Participants might experience less fatigue and clearer thinking after ketamine treatment. They could also feel better overall in terms of mood and quality of life. Since ketamine can work quickly, some people may notice improvements shortly after starting the treatment.

What are the risks? Ketamine can cause side effects like feeling dizzy, anxious, or having an unusual sense of reality (sometimes called dissociation). It may also cause temporary increases in blood pressure or heart rate. All treatments will be carefully monitored by healthcare professionals to ensure safety.

Who can participate? Adults aged 18-65 with Long COVID who have significant fatigue or thinking problems can join. People will not be able to participate if they have certain health conditions like severe heart disease, uncontrolled high blood pressure, or a history of severe mental health disorders.

Why is this study important? Long COVID affects millions of people, and many are struggling to find treatments that work. This study is one of the first to explore ketamine as a potential treatment for Long COVID symptoms. If ketamine helps, it could lead to more research and eventually new treatment options for people living with Long COVID.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years diagnosed with LC and possess a documented history of positive COVID-19 diagnostic testing or a probable infection as determined by a healthcare provider.
* One persistent symptom of fatigue or neurocognitive dysfunction as defined by rating their symptoms as moderate to severe on the screening form.
* English as a primary language OR comprehension of English suitable to understand research staff instructions.
* All participants must be eligible for MRI and will undergo MRI scans pre- and post-treatment

Exclusion Criteria:

Contraindications to ketamine therapy:

* Current substance use disorder
* Current mania or psychosis
* Recent myocardial infarction or stroke (within 1 year)
* Unstable cardiovascular disease (including uncontrolled high blood pressure > 180/110 mmHg)
* Uncontrolled seizure disorder
* Pregnancy

Additional exclusion criteria include:

* Recent COVID-19 infection or reinfection within 8 weeks
* Prior receipt of ketamine treatment
* History of treatment resistant depression (TRD) prior to development of LC

  * Defined as completing a trial (2 months of treatment at highest tolerated dose) of 3 or more psychotropic medications from at least 2 classes of medications (i.e. SSRIs, SNRIs, antipsychotic medications, or mood stabilizers such as lithium, lamotrigine, Depakote, or oxcarbazepine)
  * Psychotropic medications used during treatment of LC will not be counted as medications used for TRD
* Current severe depression or anxiety, and/or active suicidal ideation

  * Severe depression and anxiety defined as scoring > 19 on PHQ-9 screening or > 14 on GAD-7 screening.
  * Active suicidal ideation is defined as answering "yes" to question #9 on the PHQ-9
* History of bipolar disorder, schizophrenia, or schizoaffective disorder
* History of suicide attempt or psychiatric hospitalization for any reason in the last 5 years
* Current benzodiazepine or naltrexone medication use within 4 weeks of enrollment as these may decrease or block the therapeutic effect of ketamine treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
PROMIS SF v1.0 - Fatigue 8a | At enrollment and at the post-treatment assessment visit, 6 weeks following completion of the ketamine treatment.
  A patient-reported questionnaire measuring the severity and impact of fatigue on daily activities over the past 7 days. Higher scores indicate greater fatigue.
PROMIS SF v2.0 Cognitive Function 4a | At enrollment and at the post-treatment assessment visit, 6 weeks following completion of the ketamine treatment.
  A patient-reported tool that measures perceived cognitive abilities, such as memory, concentration, and mental clarity, over the past 7 days. Higher scores reflect better cognitive function.
BrainCheck Cognitive Battery | At enrollment and at the post-treatment assessment visit, 6 weeks following completion of the ketamine treatment.
  A computerized series of neuropsychological tests assessing objective cognitive functions, including memory, attention, executive function, processing speed, and response inhibition. Scores are age-normalized.
Number of participants with treatment-related adverse events as assessed by standardized interview | Adverse events will be assessed at each of the four ketamine treatment sessions and during the final post-treatment assessment, which occurs six weeks after the last ketamine injection.
  A standardized interview conducted post-treatment to identify and record any physical or psychological side effects experienced by participants during the ketamine therapy.

SECONDARY OUTCOMES:
PROMIS Global 10 v1.2 | Collected at baseline (pre-treatment) and at the post-treatment assessment (6 weeks after the final ketamine session).
  A 10-item questionnaire assessing overall physical, mental, and social health, including pain, fatigue, and emotional well-being.
NASA Task Load Index (NASA-TLX) | Collected at baseline (pre-treatment) and at the post-treatment assessment (6 weeks after the final ketamine session).
  A tool used to evaluate perceived mental workload, assessing factors like mental demand, effort, and frustration during cognitive tasks like BrainCheck.
Patient Health Questionnaire-9 (PHQ-9) | Collected before each ketamine treatment session, at baseline, and at the post-treatment assessment (6 weeks post-treatment).
  A widely used self-report measure to assess the severity of depressive symptoms over the past two weeks.
Generalized Anxiety Disorder-7 (GAD-7) | Collected before each ketamine treatment session, at baseline, and at the post-treatment assessment (6 weeks post-treatment).
  A widely used 7-item scale measuring the severity of anxiety symptoms over the past two weeks.
Depression in Medically Ill 10 Scale (DMI-10) | Collected at baseline (pre-treatment) and at the post-treatment assessment (6 weeks after the final ketamine session).
  A measure designed to assess depressive symptoms specifically in individuals with medical conditions, focusing on somatic and cognitive symptoms.
Long COVID Review of Systems | Collected at baseline (pre-treatment) and at the post-treatment assessment (6 weeks after the final ketamine session).
  A comprehensive symptom checklist adapted from the WHO's Global COVID-19 Clinical Platform, evaluating the range and severity of Long COVID symptoms.
Neuroimaging (MRI) Outcomes | Performed at baseline and repeated at the post-treatment assessment (6 weeks after the final ketamine session).
  Functional MRI (fMRI) scans will evaluate changes in brain structure and connectivity, providing insight into the neurological effects and mechanisms of ketamine.
Serum Biomarker Analysis | Collected at baseline and at the post-treatment assessment (6 weeks after the final ketamine session).
  Blood samples will be analyzed for inflammatory and metabolic markers, including cytokines and metabolites in the kynurenine pathway, to assess biological responses to ketamine treatment.

CONTACTS AND LOCATIONS:
Overall Officials: W. Michael Brode, MD, Principal Investigator — University of Texas at Austin
Locations (1):
- UT Health Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) to be shared will include de-identified data related to primary and secondary outcomes, such as patient-reported outcomes (e.g., PROMIS Fatigue and Cognitive Function scores), objective cognitive assessments from the BrainCheck battery, and adverse event reports. Additionally, de-identified neuroimaging data (for participants undergoing MRI) and biomarker data from blood samples will be included. Only data used in the results publication and relevant to the study's primary and secondary outcomes will be shared. All shared data will be stripped of personal identifiers to maintain participant confidentiality, following HIPAA guidelines.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The de-identified IPD will be made available beginning 6 months after publication of the primary study results. Data will be available for a period of 3 years following this initial release.
Access Criteria: Data will be shared with qualified researchers affiliated with academic institutions, healthcare organizations, or other research entities conducting studies related to Long COVID, neurocognitive function, or ketamine treatment. Researchers must submit a formal data request, including a summary of the proposed research and intended use of the data. Requests will be reviewed by the study's principal investigator and research team to ensure alignment with ethical guidelines and scientific merit. Approved researchers will be required to sign a data use agreement to ensure proper handling and confidentiality of the data.

REFERENCES:
- [Background] Herrera JE, Niehaus WN, Whiteson J, Azola A, Baratta JM, Fleming TK, Kim SY, Naqvi H, Sampsel S, Silver JK, Verduzco-Gutierrez M, Maley J, Herman E, Abramoff B. Multidisciplinary collaborative consensus guidance statement on the assessment and treatment of fatigue in postacute sequelae of SARS-CoV-2 infection (PASC) patients. PM R. 2021 Sep;13(9):1027-1043. doi: 10.1002/pmrj.12684. Epub 2021 Aug 24. No abstract available. PMID 34346558
- [Background] Cheng AL, Anderson J, Didehbani N, Fine JS, Fleming TK, Karnik R, Longo M, Ng R, Re'em Y, Sampsel S, Shulman J, Silver JK, Twaite J, Verduzco-Gutierrez M, Kurylo M. Multi-disciplinary collaborative consensus guidance statement on the assessment and treatment of mental health symptoms in patients with post-acute sequelae of SARS-CoV-2 infection (PASC). PM R. 2023 Dec;15(12):1588-1604. doi: 10.1002/pmrj.13085. Epub 2023 Nov 8. No abstract available. PMID 37937672
- [Background] Blitshteyn S, Whiteson JH, Abramoff B, Azola A, Bartels MN, Bhavaraju-Sanka R, Chung T, Fleming TK, Henning E, Miglis MG, Sampsel S, Silver JK, Tosto J, Verduzco-Gutierrez M, Putrino D. Multi-disciplinary collaborative consensus guidance statement on the assessment and treatment of autonomic dysfunction in patients with post-acute sequelae of SARS-CoV-2 infection (PASC). PM R. 2022 Oct;14(10):1270-1291. doi: 10.1002/pmrj.12894. Epub 2022 Oct 8. No abstract available. PMID 36169154
- [Background] Melamed E, Rydberg L, Ambrose AF, Bhavaraju-Sanka R, Fine JS, Fleming TK, Herman E, Phipps Johnson JL, Kucera JR, Longo M, Niehaus W, Oleson CV, Sampsel S, Silver JK, Smith MM, Verduzco-Gutierrez M. Multidisciplinary collaborative consensus guidance statement on the assessment and treatment of neurologic sequelae in patients with post-acute sequelae of SARS-CoV-2 infection (PASC). PM R. 2023 May;15(5):640-662. doi: 10.1002/pmrj.12976. Epub 2023 May 9. No abstract available. PMID 36989078
- [Background] Global COVID-19 Clinical Platform Case Report Form (CRF) for Post COVID condition (Post COVID-19 CRF). Accessed June 11, 2023. https://www.who.int/publications-detail-redirect/global-covid-19-clinical-platform-case-report-form-(crf)-for-post-covid-conditions-(post-covid-19-crf-)
- [Background] Valdes Hernandez Mdel C, Armitage PA, Thrippleton MJ, Chappell F, Sandeman E, Munoz Maniega S, Shuler K, Wardlaw JM. Rationale, design and methodology of the image analysis protocol for studies of patients with cerebral small vessel disease and mild stroke. Brain Behav. 2015 Nov 26;5(12):e00415. doi: 10.1002/brb3.415. eCollection 2015 Dec. PMID 26807340
- [Background] Groppell S, Soto-Ruiz KM, Flores B, Dawkins W, Smith I, Eagleman DM, Katz Y. A Rapid, Mobile Neurocognitive Screening Test to Aid in Identifying Cognitive Impairment and Dementia (BrainCheck): Cohort Study. JMIR Aging. 2019 Mar 21;2(1):e12615. doi: 10.2196/12615. PMID 31518280
- [Background] Marcantoni WS, Akoumba BS, Wassef M, Mayrand J, Lai H, Richard-Devantoy S, Beauchamp S. A systematic review and meta-analysis of the efficacy of intravenous ketamine infusion for treatment resistant depression: January 2009 - January 2019. J Affect Disord. 2020 Dec 1;277:831-841. doi: 10.1016/j.jad.2020.09.007. Epub 2020 Sep 7. PMID 33065824
- [Background] Nikolin S, Rodgers A, Schwaab A, Bahji A, Zarate C Jr, Vazquez G, Loo C. Ketamine for the treatment of major depression: a systematic review and meta-analysis. EClinicalMedicine. 2023 Aug 3;62:102127. doi: 10.1016/j.eclinm.2023.102127. eCollection 2023 Aug. PMID 37593223
- [Background] Lenze EJ, Reiersen AM, Zorumski CF, Santosh PJ. Beyond "Psychotropic": Repurposing Psychiatric Drugs for COVID-19, Alzheimer's Disease, and Cancer. J Clin Psychiatry. 2023 Mar 20;84(3):22r14494. doi: 10.4088/JCP.22r14494. PMID 36946597
- [Background] Walsh Z, Mollaahmetoglu OM, Rootman J, Golsof S, Keeler J, Marsh B, Nutt DJ, Morgan CJA. Ketamine for the treatment of mental health and substance use disorders: comprehensive systematic review. BJPsych Open. 2021 Dec 23;8(1):e19. doi: 10.1192/bjo.2021.1061. PMID 35048815
- [Background] McIntyre RS, Rosenblat JD, Nemeroff CB, Sanacora G, Murrough JW, Berk M, Brietzke E, Dodd S, Gorwood P, Ho R, Iosifescu DV, Lopez Jaramillo C, Kasper S, Kratiuk K, Lee JG, Lee Y, Lui LMW, Mansur RB, Papakostas GI, Subramaniapillai M, Thase M, Vieta E, Young AH, Zarate CA Jr, Stahl S. Synthesizing the Evidence for Ketamine and Esketamine in Treatment-Resistant Depression: An International Expert Opinion on the Available Evidence and Implementation. Am J Psychiatry. 2021 May 1;178(5):383-399. doi: 10.1176/appi.ajp.2020.20081251. Epub 2021 Mar 17. PMID 33726522
- [Background] Feder A, Parides MK, Murrough JW, Perez AM, Morgan JE, Saxena S, Kirkwood K, Aan Het Rot M, Lapidus KA, Wan LB, Iosifescu D, Charney DS. Efficacy of intravenous ketamine for treatment of chronic posttraumatic stress disorder: a randomized clinical trial. JAMA Psychiatry. 2014 Jun;71(6):681-8. doi: 10.1001/jamapsychiatry.2014.62. PMID 24740528
- [Background] Singh JB, Fedgchin M, Daly EJ, De Boer P, Cooper K, Lim P, Pinter C, Murrough JW, Sanacora G, Shelton RC, Kurian B, Winokur A, Fava M, Manji H, Drevets WC, Van Nueten L. A Double-Blind, Randomized, Placebo-Controlled, Dose-Frequency Study of Intravenous Ketamine in Patients With Treatment-Resistant Depression. Am J Psychiatry. 2016 Aug 1;173(8):816-26. doi: 10.1176/appi.ajp.2016.16010037. Epub 2016 Apr 8. PMID 27056608
- [Background] Sanacora G, Frye MA, McDonald W, Mathew SJ, Turner MS, Schatzberg AF, Summergrad P, Nemeroff CB; American Psychiatric Association (APA) Council of Research Task Force on Novel Biomarkers and Treatments. A Consensus Statement on the Use of Ketamine in the Treatment of Mood Disorders. JAMA Psychiatry. 2017 Apr 1;74(4):399-405. doi: 10.1001/jamapsychiatry.2017.0080. PMID 28249076
- [Background] McAllister-Williams RH, Arango C, Blier P, Demyttenaere K, Falkai P, Gorwood P, Hopwood M, Javed A, Kasper S, Malhi GS, Soares JC, Vieta E, Young AH, Papadopoulos A, Rush AJ. The identification, assessment and management of difficult-to-treat depression: An international consensus statement. J Affect Disord. 2020 Apr 15;267:264-282. doi: 10.1016/j.jad.2020.02.023. Epub 2020 Feb 7. PMID 32217227
- [Background] Ketamine - StatPearls - NCBI Bookshelf. Accessed March 12, 2024. https://www.ncbi.nlm.nih.gov/books/NBK470357/
- [Background] Cervia-Hasler C, Bruningk SC, Hoch T, Fan B, Muzio G, Thompson RC, Ceglarek L, Meledin R, Westermann P, Emmenegger M, Taeschler P, Zurbuchen Y, Pons M, Menges D, Ballouz T, Cervia-Hasler S, Adamo S, Merad M, Charney AW, Puhan M, Brodin P, Nilsson J, Aguzzi A, Raeber ME, Messner CB, Beckmann ND, Borgwardt K, Boyman O. Persistent complement dysregulation with signs of thromboinflammation in active Long Covid. Science. 2024 Jan 19;383(6680):eadg7942. doi: 10.1126/science.adg7942. Epub 2024 Jan 19. PMID 38236961
- [Background] Klein J, Wood J, Jaycox JR, Dhodapkar RM, Lu P, Gehlhausen JR, Tabachnikova A, Greene K, Tabacof L, Malik AA, Silva Monteiro V, Silva J, Kamath K, Zhang M, Dhal A, Ott IM, Valle G, Pena-Hernandez M, Mao T, Bhattacharjee B, Takahashi T, Lucas C, Song E, McCarthy D, Breyman E, Tosto-Mancuso J, Dai Y, Perotti E, Akduman K, Tzeng TJ, Xu L, Geraghty AC, Monje M, Yildirim I, Shon J, Medzhitov R, Lutchmansingh D, Possick JD, Kaminski N, Omer SB, Krumholz HM, Guan L, Dela Cruz CS, van Dijk D, Ring AM, Putrino D, Iwasaki A. Distinguishing features of long COVID identified through immune profiling. Nature. 2023 Nov;623(7985):139-148. doi: 10.1038/s41586-023-06651-y. Epub 2023 Sep 25. PMID 37748514
- [Background] Greene C, Connolly R, Brennan D, Laffan A, O'Keeffe E, Zaporojan L, O'Callaghan J, Thomson B, Connolly E, Argue R, Meaney JFM, Martin-Loeches I, Long A, Cheallaigh CN, Conlon N, Doherty CP, Campbell M. Blood-brain barrier disruption and sustained systemic inflammation in individuals with long COVID-associated cognitive impairment. Nat Neurosci. 2024 Mar;27(3):421-432. doi: 10.1038/s41593-024-01576-9. Epub 2024 Feb 22. PMID 38388736
- [Background] Krystal JH, Kavalali ET, Monteggia LM. Ketamine and rapid antidepressant action: new treatments and novel synaptic signaling mechanisms. Neuropsychopharmacology. 2024 Jan;49(1):41-50. doi: 10.1038/s41386-023-01629-w. Epub 2023 Jul 24. PMID 37488280
- [Background] Wong AC, Devason AS, Umana IC, Cox TO, Dohnalova L, Litichevskiy L, Perla J, Lundgren P, Etwebi Z, Izzo LT, Kim J, Tetlak M, Descamps HC, Park SL, Wisser S, McKnight AD, Pardy RD, Kim J, Blank N, Patel S, Thum K, Mason S, Beltra JC, Michieletto MF, Ngiow SF, Miller BM, Liou MJ, Madhu B, Dmitrieva-Posocco O, Huber AS, Hewins P, Petucci C, Chu CP, Baraniecki-Zwil G, Giron LB, Baxter AE, Greenplate AR, Kearns C, Montone K, Litzky LA, Feldman M, Henao-Mejia J, Striepen B, Ramage H, Jurado KA, Wellen KE, O'Doherty U, Abdel-Mohsen M, Landay AL, Keshavarzian A, Henrich TJ, Deeks SG, Peluso MJ, Meyer NJ, Wherry EJ, Abramoff BA, Cherry S, Thaiss CA, Levy M. Serotonin reduction in post-acute sequelae of viral infection. Cell. 2023 Oct 26;186(22):4851-4867.e20. doi: 10.1016/j.cell.2023.09.013. Epub 2023 Oct 16. PMID 37848036
- [Background] Leng A, Shah M, Ahmad SA, Premraj L, Wildi K, Li Bassi G, Pardo CA, Choi A, Cho SM. Pathogenesis Underlying Neurological Manifestations of Long COVID Syndrome and Potential Therapeutics. Cells. 2023 Mar 6;12(5):816. doi: 10.3390/cells12050816. PMID 36899952
- [Background] Cysique LA, Jakabek D, Bracken SG, Allen-Davidian Y, Heng B, Chow S, Dehhaghi M, Staats Pires A, Darley DR, Byrne A, Phetsouphanh C, Kelleher A, Dore GJ, Matthews GV, Guillemin GJ, Brew BJ. The kynurenine pathway relates to post-acute COVID-19 objective cognitive impairment and PASC. Ann Clin Transl Neurol. 2023 Aug;10(8):1338-1352. doi: 10.1002/acn3.51825. Epub 2023 Jun 15. PMID 37318955
- [Background] Davis HE, McCorkell L, Vogel JM, Topol EJ. Long COVID: major findings, mechanisms and recommendations. Nat Rev Microbiol. 2023 Mar;21(3):133-146. doi: 10.1038/s41579-022-00846-2. Epub 2023 Jan 13. PMID 36639608
- [Background] Davis HE, Assaf GS, McCorkell L, Wei H, Low RJ, Re'em Y, Redfield S, Austin JP, Akrami A. Characterizing long COVID in an international cohort: 7 months of symptoms and their impact. EClinicalMedicine. 2021 Aug;38:101019. doi: 10.1016/j.eclinm.2021.101019. Epub 2021 Jul 15. PMID 34308300
- [Background] Thaweethai T, Jolley SE, Karlson EW, Levitan EB, Levy B, McComsey GA, McCorkell L, Nadkarni GN, Parthasarathy S, Singh U, Walker TA, Selvaggi CA, Shinnick DJ, Schulte CCM, Atchley-Challenner R, Alba GA, Alicic R, Altman N, Anglin K, Argueta U, Ashktorab H, Baslet G, Bassett IV, Bateman L, Bedi B, Bhattacharyya S, Bind MA, Blomkalns AL, Bonilla H, Brim H, Bush PA, Castro M, Chan J, Charney AW, Chen P, Chibnik LB, Chu HY, Clifton RG, Costantine MM, Cribbs SK, Davila Nieves SI, Deeks SG, Duven A, Emery IF, Erdmann N, Erlandson KM, Ernst KC, Farah-Abraham R, Farner CE, Feuerriegel EM, Fleurimont J, Fonseca V, Franko N, Gainer V, Gander JC, Gardner EM, Geng LN, Gibson KS, Go M, Goldman JD, Grebe H, Greenway FL, Habli M, Hafner J, Han JE, Hanson KA, Heath J, Hernandez C, Hess R, Hodder SL, Hoffman MK, Hoover SE, Huang B, Hughes BL, Jagannathan P, John J, Jordan MR, Katz SD, Kaufman ES, Kelly JD, Kelly SW, Kemp MM, Kirwan JP, Klein JD, Knox KS, Krishnan JA, Kumar A, Laiyemo AO, Lambert AA, Lanca M, Lee-Iannotti JK, Logarbo BP, Longo MT, Luciano CA, Lutrick K, Maley JH, Mallett G, Marathe JG, Marconi V, Marshall GD, Martin CF, Matusov Y, Mehari A, Mendez-Figueroa H, Mermelstein R, Metz TD, Morse R, Mosier J, Mouchati C, Mullington J, Murphy SN, Neuman RB, Nikolich JZ, Ofotokun I, Ojemakinde E, Palatnik A, Palomares K, Parimon T, Parry S, Patterson JE, Patterson TF, Patzer RE, Peluso MJ, Pemu P, Pettker CM, Plunkett BA, Pogreba-Brown K, Poppas A, Quigley JG, Reddy U, Reece R, Reeder H, Reeves WB, Reiman EM, Rischard F, Rosand J, Rouse DJ, Ruff A, Saade G, Sandoval GJ, Santana JL, Schlater SM, Sciurba FC, Shepherd F, Sherif ZA, Simhan H, Singer NG, Skupski DW, Sowles A, Sparks JA, Sukhera FI, Taylor BS, Teunis L, Thomas RJ, Thorp JM, Thuluvath P, Ticotsky A, Tita AT, Tuttle KR, Urdaneta AE, Valdivieso D, VanWagoner TM, Vasey A, Verduzco-Gutierrez M, Wallace ZS, Ward HD, Warren DE, Weiner SJ, Welch S, Whiteheart SW, Wiley Z, Wisnivesky JP, Yee LM, Zisis S, Horwitz LI, Foulkes AS; RECOVER Consortium. Development of a Definition of Postacute Sequelae of SARS-CoV-2 Infection. JAMA. 2023 Jun 13;329(22):1934-1946. doi: 10.1001/jama.2023.8823. PMID 37278994
- [Background] Perlis RH, Santillana M, Ognyanova K, Safarpour A, Lunz Trujillo K, Simonson MD, Green J, Quintana A, Druckman J, Baum MA, Lazer D. Prevalence and Correlates of Long COVID Symptoms Among US Adults. JAMA Netw Open. 2022 Oct 3;5(10):e2238804. doi: 10.1001/jamanetworkopen.2022.38804. PMID 36301542
- [Background] Logue JK, Franko NM, McCulloch DJ, McDonald D, Magedson A, Wolf CR, Chu HY. Sequelae in Adults at 6 Months After COVID-19 Infection. JAMA Netw Open. 2021 Feb 1;4(2):e210830. doi: 10.1001/jamanetworkopen.2021.0830. PMID 33606031
- [Background] Bull-Otterson L, Baca S, Saydah S, et al. Post-COVID Conditions Among Adult COVID-19 Survivors Aged 18-64 and ≥65 Years - United States, March 2020-November 2021. MMWR Morb Mortal Wkly Rep. 2022;71(21):713-717. doi:10.15585/mmwr.mm7121e1
- [Background] CDC. Post-COVID Conditions. Centers for Disease Control and Prevention. Published September 1, 2022. Accessed December 6, 2022. https://www.cdc.gov/coronavirus/2019-ncov/long-term-effects/index.html
- [Result] Chakraborty C, Bhattacharya M. The current landscape of long COVID clinical trials: NIH's RECOVER to Stanford Medicine's STOP-PASC initiative. Mol Ther Nucleic Acids. 2023 Aug 28;33:887-889. doi: 10.1016/j.omtn.2023.08.016. eCollection 2023 Sep 12. No abstract available. PMID 37680987
- [Result] Fazekas F, Chawluk JB, Alavi A, Hurtig HI, Zimmerman RA. MR signal abnormalities at 1.5 T in Alzheimer's dementia and normal aging. AJR Am J Roentgenol. 1987 Aug;149(2):351-6. doi: 10.2214/ajr.149.2.351. PMID 3496763
- [Result] Nikolich JZ, Rosen CJ. Toward Comprehensive Care for Long Covid. N Engl J Med. 2023 Jun 8;388(23):2113-2115. doi: 10.1056/NEJMp2304550. Epub 2023 May 9. No abstract available. PMID 37158440
- [Result] Kopra E, Mondelli V, Pariante C, Nikkheslat N. Ketamine's effect on inflammation and kynurenine pathway in depression: A systematic review. J Psychopharmacol. 2021 Aug;35(8):934-945. doi: 10.1177/02698811211026426. Epub 2021 Jun 26. PMID 34180293
- [Result] Lullau APM, Haga EMW, Ronold EH, Dwyer GE. Antidepressant mechanisms of ketamine: a review of actions with relevance to treatment-resistance and neuroprogression. Front Neurosci. 2023 Aug 8;17:1223145. doi: 10.3389/fnins.2023.1223145. eCollection 2023. PMID 37614344
- [Result] Kang MJY, Hawken E, Vazquez GH. The Mechanisms Behind Rapid Antidepressant Effects of Ketamine: A Systematic Review With a Focus on Molecular Neuroplasticity. Front Psychiatry. 2022 Apr 25;13:860882. doi: 10.3389/fpsyt.2022.860882. eCollection 2022. PMID 35546951
- [Result] Meier TB, Savitz J. The Kynurenine Pathway in Traumatic Brain Injury: Implications for Psychiatric Outcomes. Biol Psychiatry. 2022 Mar 1;91(5):449-458. doi: 10.1016/j.biopsych.2021.05.021. Epub 2021 May 31. PMID 34266671
- [Result] Al-Aly Z, Topol E. Solving the puzzle of Long Covid. Science. 2024 Feb 23;383(6685):830-832. doi: 10.1126/science.adl0867. Epub 2024 Feb 22. PMID 38386747
- [Result] Aziz R, Siles N, Kelley M, Wylie D, Melamed E, Brode WM. Clinical characteristics of Long COVID patients presenting to a dedicated academic post-COVID-19 clinic in Central Texas. Sci Rep. 2023 Dec 11;13(1):21971. doi: 10.1038/s41598-023-48502-w. PMID 38081885
- [Result] Xie Y, Bowe B, Al-Aly Z. Burdens of post-acute sequelae of COVID-19 by severity of acute infection, demographics and health status. Nat Commun. 2021 Nov 12;12(1):6571. doi: 10.1038/s41467-021-26513-3. PMID 34772922